CLINICAL TRIAL: NCT00396981
Title: A Prospective, Randomized, Multicenter Trial Investigating Matrix 2® and GDC® Detachable Coils for the Treatment of Intracranial Saccular Aneurysms
Brief Title: MAPS Trial: Matrix And Platinum Science
Acronym: MAPS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stryker Neurovascular (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: T4902; BSC0015 (Other: Stryker Neurovascular)
Record Dates: First submitted 2006-11-06; First posted 2006-11-08 (Estimated); Results first posted 2014-03-18 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-01

CONDITIONS: Intracranial Aneurysms
Keywords: Intracranial saccular aneurysms; Endovascular coiling therapy; Retreatment; Raymond scale; Matrix; GDC; Guglielmi Detachable Coil
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Matrix 2® Coils (Active Comparator): Matrix 2® Coils for endovascular aneurysm occlusion
  Interventions: Device: Matrix 2® coils for endovascular aneurysm occlusion
- GDC® Coils (Active Comparator): GDC® Coils for endovascular aneurysm occlusion
  Interventions: Device: GDC® coils for endovascular aneurysm occlusion

INTERVENTIONS:
Device: Matrix 2® coils for endovascular aneurysm occlusion — endovascular aneurysm occlusion coil
  Arms: Matrix 2® Coils
Device: GDC® coils for endovascular aneurysm occlusion — endovascular aneurysm occlusion coil
  Arms: GDC® Coils

SUMMARY:
Primary Objectives:

* To establish Target Aneurysm Recurrence (TAR) rates for Matrix 2® and GDC® Coils used for the treatment of intracranial saccular aneurysms. TAR is defined as clinically relevant recurrence resulting in: target aneurysm reintervention, rupture/re-rupture and/or death from an unknown cause.
* To correlate defined angiographic endpoints with TAR rates and assess their predictive value, thereby providing a framework to establish clinically relevant endpoints for future studies.

Secondary Objectives:

* To evaluate device characteristics, incidence and severity of device-related adverse events, including death, neurological deterioration and changes in functional abilities.
* To establish angiographic recurrence rates for Matrix 2® and GDC® Coils used for the treatment of intracranial saccular aneurysms.
* To explore an experimental, quantitative and volumetric endpoint and correlate these with existing qualitative assessments.

DETAILED DESCRIPTION:
The endovascular treatment of intracranial aneurysms has become an accepted alternative to surgical repair given the many recent advances with neurointerventional devices and procedures. The introduction of GDC coils in 1993 provided physicians and their patients a less invasive treatment option. Additionally, the results of two large international trials, ISAT and ISUIA, have shown the benefits of endovascular treatment over surgery for treatment of specific types of aneurysms. One limitation of endovascular coil embolization is aneurysm recurrence or recanalization which is not infrequently observed angiographically at follow up. Aneurysm recanalization may be a result of aneurysm morphology, anatomic location and flow orientation, aneurysm regrowth or the degree of coil compaction. Despite the widespread adoption of endovascular aneurysm coiling, there remains much to be learned about the efficacy and optimization of this treatment modality.

The goal of endovascular embolization of intracranial aneurysms is to prevent rupture or re-rupture. Fortunately, the incidence of aneurysm rupture following coil embolization is very low. Follow-up angiographic analysis to evaluate the occlusion and stability of the treated aneurysm provides a surrogate endpoint against which to weigh the likelihood of rupture/re-rupture. However, angiographic interpretation is subjective, operator dependent and can be influenced by multiple confounding variables.

The MAPS trial will examine Target Aneurysm Recurrence Rates: clinically relevant recurrence rates resulting in target aneurysm reintervention, rupture/re-rupture and/or death from an unknown cause for Matrix 2® and GDC® Coils used for the treatment of intracranial saccular aneurysms. The trial will compare TAR rates to recurrences measured by angiographic analysis and assess the utility of angiographic analysis for predicting clinically relevant recurrences.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is between 18 and 80 years of age (inclusive).
2. Patient has a documented untreated intracranial saccular aneurysm 4-20 mm diameter angiographic lumen, ruptured or unruptured, suitable for embolization with coils.
3. Both GDC® Coils and Matrix 2® Coils (Every attempt should be made to treat with as much randomized coil type as possible to achieve optimal occlusion.) are treatment options (all shapes allowed with exception of GDC VortX Coil).
4. Target aneurysm can be adequately coiled at index procedure (NO staged coiling procedures). If a Neuroform stent is to be placed during a separate preliminary procedure, then screening and enrollment for the coiling procedure must take place after the stenting procedure is completed.
5. Target aneurysm morphology allows for adequate retention of coils within the aneurysmal sac without occlusion of the parent artery, as determined by the treating physician.
6. Patient (or patient's legally authorized representative for centers in the United States) has provided written informed consent.
7. Patient is willing and able to comply with protocol follow-up requirements.

Exclusion Criteria:

1. Patient is < 18 or > 80 years old.
2. Target aneurysm is not saccular in nature (mycotic, fusiform, dissecting).
3. Target aneurysm is > 20 mm maximum luminal dimension, < 4 mm maximum luminal dimension.
4. Target aneurysm has been previously treated by surgery or endovascular therapy.
5. Target aneurysm is in the physician's estimation unlikely to be successfully treated by endovascular techniques.
6. Patient presents as Hunt and Hess grade IV or V for a ruptured aneurysm.
7. Patient presents with Modified Rankin Score 4 or 5 at baseline.
8. Patient is concurrently enrolled in another investigational drug or device study unless permission is granted by the sponsor.
9. Patient has known hypersensitivity to Polyglycolic Polylactic Acid (PGLA), platinum, nickel, stainless steel or structurally related compounds found in Matrix 2® Coils and/or GDC® Coils.
10. Patients who have had or could have a severe reaction to contrast agents that cannot be adequately pre-medicated prior to the coiling procedure.
11. Patients who are unable to complete scheduled follow up assessments at the enrolling center due to limited life expectancy (< 12 months), comorbidities or geographical considerations.
12. Planned use of adjunctive therapy stents except Neuroform is not allowed.
13. Patients with Moya-Moya disease, AVMs, AV fistula, intracranial tumors, intracranial hematoma (unrelated to target aneurysm), significant atherosclerotic stenosis, tortuousity or other conditions preventing access to the target aneurysm.
14. Patients with multiple aneurysms.
15. Target aneurysm with significant thrombosis that may increase the likelihood of recanalization at the discretion of the investigator.
16. Female patient has a positive pregnancy assessment at baseline.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 626 (Actual)
Dates: Start 2007-03; Primary Completion 2011-01 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: S. Claiborne Johnston, MD, PhD, Principal Investigator — University of California, San Francisco, CA; Cameron McDougall, MD, Principal Investigator — Barrow Neurological Institute, Phoenix, AZ; Anil Gholkar, MD, Principal Investigator — Newcastle Upon Tyne Hospitals, NHS Trust, UK
Locations (43):
- United States (26):
  - St. Joseph's Hospital Barrow Neurological Institute, Phoenix, Arizona
  - Tucson Medical Center, Tucson, Arizona
  - Yale-New Haven Hospital, New Haven, Connecticut
  - Rush Presbyterian, Chicago, Illinois
  - The Universtiy of Iowa, Iowa City, Iowa
  - University of Maryland, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Massachusetts Worcester, Worcester, Massachusetts
  - Providence Detroit, Southfield, Michigan
  - St. Joseph's Hospital, Saint Paul, Minnesota
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Barnes Jewish Mallinckrodt Institute of Radiology, St Louis, Missouri
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - University of New Mexico Department of Neurosurgery, Albuquerque, New Mexico
  - Stony Brook Medical Center, Stony Brook, New York
  - Carolina Neurosurgery & Spine Associates, PA, Charlotte, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Mercy Health Center, Oklahoma City, Oklahoma
  - OHSU, Portland, Oregon
  - Medical University of South Carolina, Charleston, South Carolina
  - Fort Sanders Regional Medical Center, Knoxville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Methodist Hospital, Houston, Texas
  - University of Washington Harborview Medical Center, Seattle, Washington
  - Sacred Heart Providence, Spokane, Washington
  - University of Wisconsin Hospital and Center, Madison, Wisconsin
- Royal Melbourne Hospital, Parkville, Australia
- Montreal Neurological Institute and Hospital, Montreal, Quebec, Canada
- Xuan Wu Hospital, Beijing, China
- CHU Montpelier, Montpellier, France
- Germany (4):
  - Klinikum Augsburg, Augsburg
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau
  - Asklepios Klinik Altona, Hamburg
  - Universitaetsklinikum des Saarlandes, Homburg/Saar
- Instituto Nacional de Neurologia e Neurocirurgia, Mexico City, Mexico City, Mexico
- Rikshospitalet University Hospital, Oslo, Norway
- Spain (4):
  - Hospital General, Alicante
  - Hospital Clinico Y provincial, Barcelona
  - Hospital Donostia, Donostia / San Sebastian
  - Clinica Ntra Sra Del Rosario Hospital Ruber Internacional, Madrid
- Istanbul University Cerrahpaşa Tıp Fakültesi, Kocamustafapaşa, Istanbul, Turkey (Türkiye)
- United Kingdom (2):
  - The Walton Centre, Fazakerley, Liverpool
  - Newcastle General Hospital Department of Neuroradiology, Tyne and Wear

REFERENCES:
- [Derived] McDougall CG, Johnston SC, Gholkar A, Barnwell SL, Vazquez Suarez JC, Masso Romero J, Chaloupka JC, Bonafe A, Wakhloo AK, Tampieri D, Dowd CF, Fox AJ, Imm SJ, Carroll K, Turk AS; MAPS Investigators. Bioactive versus bare platinum coils in the treatment of intracranial aneurysms: the MAPS (Matrix and Platinum Science) trial. AJNR Am J Neuroradiol. 2014 May;35(5):935-42. doi: 10.3174/ajnr.A3857. Epub 2014 Jan 30. PMID 24481333
- [Derived] Hetts SW, Turk A, English JD, Dowd CF, Mocco J, Prestigiacomo C, Nesbit G, Ge SG, Jin JN, Carroll K, Murayama Y, Gholkar A, Barnwell S, Lopes D, Johnston SC, McDougall C; Matrix and Platinum Science Trial Investigators. Stent-assisted coiling versus coiling alone in unruptured intracranial aneurysms in the matrix and platinum science trial: safety, efficacy, and mid-term outcomes. AJNR Am J Neuroradiol. 2014 Apr;35(4):698-705. doi: 10.3174/ajnr.A3755. Epub 2013 Nov 1. PMID 24184523

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment in the study occurred over 31 months at 26 sites in the US and 17 International. Each site was allowed to enroll up to 60 consecutive subjects; recruitment for the study was competitive. The first subject was enrolled on 29 March 2007 and the enrollment completed on 21 October 2009. A total of 626 subjects were enrolled.
Groups:
- Matrix 2® Coils for Endovascular Aneurysm Occlusion: Matrix 2® Coils for endovascular aneurysm occlusion
  Matrix 2® coils for endovascular aneurysm occlusion : endovascular aneurysm occlusion coil
- GDC® Coils for Endovascular Aneurysm Occlusion: GDC® Coils for endovascular aneurysm occlusion
  GDC® coils for endovascular aneurysm occlusion : endovascular aneurysm occlusion coil
Period: Overall Study
Arm/Group | Matrix 2® Coils for Endovascular Aneurysm Occlusion | GDC® Coils for Endovascular Aneurysm Occlusion
Started | 311 | 315
Completed | 296 | 306
Not Completed | 15 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Matrix 2® Coils for Endovascular Aneurysm Occlusion | GDC® Coils for Endovascular Aneurysm Occlusion | Total
Number analyzed (Participants) | 311 | 315 | 626
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.7 (11.6) | 54.4 (13.2) | 55.0 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 229 | 211 | 440
  Male | 82 | 104 | 186
Region of Enrollment [Number; unit: participants]
  France | 17 | 15 | 32
  United States | 183 | 190 | 373
  Mexico | 1 | 2 | 3
  Canada | 16 | 15 | 31
  Spain | 46 | 44 | 90
  Turkey | 4 | 6 | 10
  Australia | 1 | 3 | 4
  Norway | 6 | 5 | 11
  Germany | 13 | 10 | 23
  China | 7 | 9 | 16
  United Kingdom | 17 | 16 | 33

OUTCOME MEASURES:

1. Primary Outcome: Target Aneurysm Recurrence (TAR) Defined as Clinically Relevant Recurrence Resulting in Target Aneurysm Reintervention, Rupture/Re-rupture and/or Death From an Unknown Cause.
Time Frame: 12 months
Population: A totoal of 630 subjects were planned for the study. All enrolled MAPS trial subjects' data is included in the ITT anaylsis except for four subjects who were excluded due to the following reasons: one subject did not have an aneurysm and three subjects', a the request of the IRB, due to non GCP compliance in obtaining the inofrmed consent.
Measure: Number; unit: participants
Groups:
- Matrix Coils: Matrix 2® Coils for endovascular aneurysm occlusion
- GDC Coils: GDC® Coils for endovascular aneurysm occlusion
Arm/Group | Matrix Coils | GDC Coils
Number analyzed (Participants) | 311 | 315
participants | 34 | 35
Statistical Analysis 1: Comparison: Matrix Coils; Intent-to-Treat, All Subjects (N=626) GDC (N=315) Matrix (N=311) All Subjects (N=626) Subjects Who Met Primary Endpoint 35 (11.1%) 34 (10.9%) 69 (11.0%); Test type: Non-Inferiority or Equivalence — This study used a non-inferiority design to demonstrate that the Matrix Coil is non-inferior to the GDC Coil, with a clinically acceptable non-inferiority margin set at 10%. Non-inferiority was used to establish the baseline estimate, which future superiority studies could be conducted. Non-inferiority was shown with a one-sided 95% CI of the difference less than the pre-specified 10% margin; p = 0.76, Log Rank

2. Secondary Outcome: Angiographic Assessments
Description: Number of participants with angiographic assessment of "complete obliteration".
Time Frame: Reintervention or 12 months
Measure: Number; unit: participants
Arm/Group | Matrix Coils | GDC Coils
Number analyzed (Participants) | 238 | 250
participants | 87 | 89

3. Secondary Outcome: Neurological Assessments
Description: The changes in modified Rankin Scores from pre-procedure to 12-month were measured. the outcome below reflects "same or better".
Time Frame: 12 months
Measure: Number; unit: percentage of participants
Arm/Group | Matrix Coils | GDC Coils
Number analyzed (Participants) | 311 | 315
percentage of participants | 90.1 | 88.3

4. Secondary Outcome: Technical Procedure Success
Time Frame: Post-procedure
Measure: Number; unit: percentage of participants
Arm/Group | Matrix Coils | GDC Coils
Number analyzed (Participants) | 311 | 315
percentage of participants | 96.8 | 97.5

5. Secondary Outcome: Target Aneurysm Recurrence
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Matrix Coils | GDC Coils
Number analyzed (Participants) | 311 | 315
participants | 42 | 42

6. Secondary Outcome: Target Aneurysm Recurrence
Time Frame: 3 years
Measure: Number; unit: participants
Arm/Group | Matrix Coils | GDC Coils
Number analyzed (Participants) | 311 | 315
participants | 43 | 45

7. Secondary Outcome: Target Aneurysm Recurrence
Time Frame: 5 years
Measure: Number; unit: participants
Arm/Group | Matrix Coils | GDC Coils
Number analyzed (Participants) | 311 | 315
participants | 44 | 46

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Matrix Coils | GDC Coils
Serious Adverse Events (participants affected / at risk) | 85/311 | 80/315
Other Adverse Events (participants affected / at risk) | 112/311 | 120/315
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Matrix Coils (N=311) | GDC Coils (N=315)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Total (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac valve disease (Cardiac disorders) | 1 (1) | 0 (0)
Cardiovascular disorder (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0)
Total (Cardiac disorders) | 7 (8) | 5 (5)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Total (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 1 (1) | 0 (0)
Total (Eye disorders) | 1 (1) | 0 (0)
Diverticular perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Peritonitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Total (Gastrointestinal disorders) | 3 (3) | 4 (4)
Catheter site discharge (General disorders) | 0 (0) | 1 (1)
Catheter site haematoma (General disorders) | 2 (2) | 2 (2)
Catheter site haemorrhage (General disorders) | 2 (2) | 0 (0)
Death (General disorders) | 3 (3) | 0 (0)
Multi-organ failure (General disorders) | 1 (1) | 0 (0)
Total (General disorders) | 8 (8) | 3 (3)
Chronic hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Total (Hepatobiliary disorders) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Total (Immune system disorders) | 0 (0) | 1 (1)
Arthritis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Central nervous system infection (Infections and infestations) | 2 (2) | 0 (0)
Clostridial infection (Infections and infestations) | 1 (2) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Meningitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3) | 2 (2)
Pneumonia escherichia (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (3) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Total (Infections and infestations) | 11 (14) | 5 (5)
Brain herniation (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Total (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Blood pressure increased (Investigations) | 0 (0) | 1 (1)
Sputum culture positive (Investigations) | 1 (1) | 0 (0)
Total (Investigations) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Total (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Total (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Benign cardiac neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Total (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Autonomic nervous system imbalance (Nervous system disorders) | 0 (0) | 1 (1)
Basilar artery thrombosis (Nervous system disorders) | 1 (1) | 0 (0)
Brain oedema (Nervous system disorders) | 2 (2) | 1 (1)
Carotid arterial embolus (Nervous system disorders) | 1 (1) | 0 (0)
Carotid artery dissection (Nervous system disorders) | 2 (2) | 2 (2)
Carotid artery thrombosis (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral artery embolism (Nervous system disorders) | 1 (1) | 2 (2)
Cerebral artery thrombosis (Nervous system disorders) | 9 (9) | 8 (8)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (1)
Diplegia (Nervous system disorders) | 1 (1) | 0 (0)
Embolic stroke (Nervous system disorders) | 1 (1) | 2 (2)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 3 (3) | 3 (3)
Headache (Nervous system disorders) | 2 (2) | 6 (6)
Hemiparesis (Nervous system disorders) | 0 (0) | 1 (1)
Hydrocephalus (Nervous system disorders) | 3 (3) | 6 (6)
IIIrd nerve disorder (Nervous system disorders) | 0 (0) | 1 (1)
Intracranial aneurysm (Nervous system disorders) | 0 (0) | 1 (1)
Intracranial pressure increased (Nervous system disorders) | 1 (1) | 4 (4)
Ischaemic neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 16 (16) | 14 (15)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1)
Nervous system disorder (Nervous system disorders) | 0 (0) | 1 (1)
Neurological symptom (Nervous system disorders) | 1 (1) | 0 (0)
Paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Ruptured cerebral aneurysm (Nervous system disorders) | 8 (8) | 9 (9)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 4 (4) | 3 (3)
Total (Nervous system disorders) | 52 (64) | 53 (69)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Total (Psychiatric disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Total (Renal and urinary disorders) | 0 (0) | 1 (1)
Cervical dysplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Total (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cryptogenic organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Total (Respiratory, thoracic and mediastinal disorders) | 6 (8) | 6 (6)
Artery dissection (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Femoral artery aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Femoral artery occlusion (Vascular disorders) | 0 (0) | 1 (1)
Iliac artery stenosis (Vascular disorders) | 0 (0) | 1 (1)
Peripheral vascular disorder (Vascular disorders) | 1 (1) | 0 (0)
Thrombophlebitis superficial (Vascular disorders) | 1 (1) | 0 (0)
Vascular pseudoaneurysm (Vascular disorders) | 2 (2) | 1 (1)
Vasospasm (Vascular disorders) | 18 (19) | 20 (29)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 1 (1)
Vessel perforation (Vascular disorders) | 1 (1) | 1 (1)
Total (Vascular disorders) | 24 (27) | 24 (34)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Matrix Coils (N=311) | GDC Coils (N=315)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 2 (2)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Total (Blood and lymphatic system disorders) | 3 (3) | 3 (3)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Arrhythmia supraventricular (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 2 (2)
Cardiac failure congestive (Cardiac disorders) | 2 (2) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 3 (3) | 2 (2)
Total (Cardiac disorders) | 7 (8) | 7 (7)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Total (Ear and labyrinth disorders) | 2 (2) | 1 (1)
Diabetes insipidus (Endocrine disorders) | 0 (0) | 1 (1)
Total (Endocrine disorders) | 0 (0) | 1 (1)
Blindness unilateral (Eye disorders) | 0 (0) | 1 (1)
Diplopia (Eye disorders) | 3 (3) | 1 (1)
Eye pain (Eye disorders) | 1 (1) | 2 (2)
Eye swelling (Eye disorders) | 1 (1) | 0 (0)
Macular degeneration (Eye disorders) | 0 (0) | 1 (1)
Photophobia (Eye disorders) | 1 (1) | 0 (0)
Photopsia (Eye disorders) | 1 (1) | 0 (0)
Retinal artery occlusion (Eye disorders) | 0 (0) | 1 (1)
Retinal haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Strabismus (Eye disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 3 (3) | 4 (4)
Visual disturbance (Eye disorders) | 1 (1) | 5 (5)
Vitreous floaters (Eye disorders) | 0 (0) | 1 (1)
Total (Eye disorders) | 10 (13) | 15 (16)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hernial eventration (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 10 (10) | 10 (10)
Tongue disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (4) | 3 (3)
Total (Gastrointestinal disorders) | 14 (20) | 13 (16)
Adverse drug reaction (General disorders) | 2 (2) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1)
Catheter site discharge (General disorders) | 6 (6) | 10 (10)
Catheter site haematoma (General disorders) | 12 (12) | 16 (16)
Catheter site haemorrhage (General disorders) | 4 (4) | 3 (3)
Catheter site pain (General disorders) | 8 (8) | 6 (6)
Catheter site rash (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 2 (2)
Fatigue (General disorders) | 1 (1) | 0 (0)
Hyperthermia (General disorders) | 1 (1) | 0 (0)
Infusion site extravasation (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Peripheral coldness (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 4 (4) | 2 (2)
Total (General disorders) | 33 (43) | 31 (40)
Contrast media allergy (Immune system disorders) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Total (Immune system disorders) | 0 (0) | 3 (3)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Catheter site infection (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 1 (1) | 0 (0)
Hepatitis E (Infections and infestations) | 1 (1) | 0 (0)
Infusion site infection (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 2 (2)
Meningitis (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 5 (5) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Tracheitis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection bact (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 8 (9) | 9 (9)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Total (Infections and infestations) | 21 (25) | 15 (18)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Patella fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural hypertension (Injury, poisoning and procedural complications) | 1 (1) | 4 (4)
Procedural hypotension (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural nausea (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radiation skin injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Scratch (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skeletal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Total (Injury, poisoning and procedural complications) | 5 (5) | 10 (10)
Electrocardiogram ST segment abnormal (Investigations) | 1 (1) | 0 (0)
Troponin increased (Investigations) | 0 (0) | 1 (1)
Ultrasound Doppler abnormal (Investigations) | 0 (0) | 1 (1)
Urine sodium increased (Investigations) | 0 (0) | 1 (1)
Total (Investigations) | 1 (1) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperchloraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (4) | 2 (2)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Metabolic disorder (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Total (Metabolism and nutrition disorders) | 7 (12) | 7 (13)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Total (Musculoskeletal and connective tissue disorders) | 5 (6) | 13 (14)
Balance disorder (Nervous system disorders) | 2 (2) | 1 (1)
Brain oedema (Nervous system disorders) | 0 (0) | 1 (1)
CNS ventriculitis (Nervous system disorders) | 0 (0) | 1 (1)
Carotid artery dissection (Nervous system disorders) | 1 (1) | 1 (1)
Carotid artery thrombosis (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral artery embolism (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral artery occlusion (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral artery stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral artery thrombosis (Nervous system disorders) | 7 (7) | 2 (2)
Convulsion (Nervous system disorders) | 0 (0) | 2 (2)
Coordination abnormal (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 3 (3) | 1 (1)
Embolic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 54 (59) | 57 (68)
Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 3 (3)
Intracranial aneurysm (Nervous system disorders) | 2 (2) | 0 (0)
Intracranial pressure increased (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 3 (3) | 3 (3)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 1 (1) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Peroneal nerve palsy (Nervous system disorders) | 0 (0) | 1 (1)
Ruptured cerebral aneurysm (Nervous system disorders) | 1 (1) | 1 (1)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1)
Sensory loss (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 2 (2) | 4 (5)
Tremor (Nervous system disorders) | 2 (2) | 0 (0)
VIth nerve paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Total (Nervous system disorders) | 73 (89) | 78 (100)
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 1 (1)
Sleep disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Total (Psychiatric disorders) | 7 (7) | 4 (4)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Urethral haemorrhage (Renal and urinary disorders) | 0 (0) | 2 (2)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Total (Renal and urinary disorders) | 0 (0) | 4 (4)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Total (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 7 (8)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (4) | 4 (4)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Increased tendency to bruise (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Rash generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Total (Skin and subcutaneous tissue disorders) | 6 (6) | 9 (9)
Artery dissection (Vascular disorders) | 1 (1) | 1 (1)
Blood pressure fluctuation (Vascular disorders) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 3 (3) | 0 (0)
Hypotension (Vascular disorders) | 6 (6) | 7 (7)
Intermittent claudication (Vascular disorders) | 1 (1) | 0 (0)
Peripheral artery aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0)
Vasospasm (Vascular disorders) | 9 (9) | 8 (8)
Total (Vascular disorders) | 23 (23) | 17 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less